CLINICAL TRIAL: NCT03784677
Title: A Phase I Study of SOR-C13 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0680; NCI-2018-02835 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0680 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-12-18; First posted 2018-12-24 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Advanced Malignant Solid Neoplasm; Refractory Malignant Solid Neoplasm; Refractory Ovarian Carcinoma; Refractory Pancreatic Carcinoma; Stage II Pancreatic Cancer AJCC v8; Stage IIA Pancreatic Cancer AJCC v8; Stage IIB Pancreatic Cancer AJCC v8; Stage III Ovarian Cancer AJCC v8; Stage III Pancreatic Cancer AJCC v8; Stage III Prostate Cancer AJCC v8; Stage IIIA Ovarian Cancer AJCC v8; Stage IIIA Prostate Cancer AJCC v8; Stage IIIB Ovarian Cancer AJCC v8; Stage IIIB Prostate Cancer AJCC v8; Stage IIIC Ovarian Cancer AJCC v8; Stage IIIC Prostate Cancer AJCC v8; Stage IV Ovarian Cancer AJCC v8; Stage IV Pancreatic Cancer AJCC v8; Stage IV Prostate Cancer AJCC v8; Stage IVA Ovarian Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8; Stage IVB Ovarian Cancer AJCC v8; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Ovarian Neoplasms; Pancreatic Neoplasms; Prostatic Neoplasms | interventions — SOR-C13

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (TRPV6 calcium channel inhibitor SOR-C13) (Experimental): Patients receive TRPV6 calcium channel inhibitor SOR-C13 IV over 2 hours on days 1, 2, 8, 9, 15, 16, 22, and 23. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: TRPV6 Calcium Channel Inhibitor SOR-C13

INTERVENTIONS:
Drug: TRPV6 Calcium Channel Inhibitor SOR-C13 — Given IV
  Other Names: SOR-C13

SUMMARY:
This phase I trial studies the side effects and best dose of SOR-C13 in treating patients with solid tumors that have spread to other places in the body (advanced) and does not respond to treatment. Drugs used in chemotherapy, such as SOR-C13, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To define the maximum tolerated doses (MTD) of TRPV6 calcium channel inhibitor SOR-C13 (SOR-C13) in subjects with advanced solid tumor cancers of epithelial origin.

II. To define the safety profiles of the treatment.

SECONDARY OBJECTIVES:

I. To evaluate clinical response signals to the treatment. II. To assess predictive biomarkers (baseline molecular mutation status) and/or resistant pathways by comparing molecular signatures at baseline versus at time of relapse in patients who have achieved objective responses.

OUTLINE: This is a dose-escalation study.

Patients receive TRPV6 calcium channel inhibitor SOR-C13 intravenously (IV) over 2 hours on days 1, 2, 8, 9, 15, 16, 22, and 23. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for this trial, patients must meet all of the following eligibility criteria.

1. Subjects with a histologic diagnosis of solid tumor cancers of epithelial origin (metastatic epithelial ovarian, pancreatic and prostate cancers are preferred since these tumor types have TRPV6 overexpression).
2. Subjects with advanced refractory cancer for which standard curative or palliative measures do not exist or are no longer effective. There is no limitation on the number or types of prior therapy.
3. Patients must have measurable or evaluable disease, as defined by Response Evaluation Criteria in Solid Tumors 1.1 (RECIST1.1).
4. Men or women aged ≥ 18 years.
5. Women of child-bearing potential (who are not postmenopausal for at least one year or are not surgically sterile) and men must agree to use adequate contraception (e.g., hormonal, barrier device, or abstinence) prior to study entry, for the duration of study participation, and for 30 days after the last dose the study agents.
6. Patients must have an ECOG performance status of 0 to 1.
7. Patients must have adequate organ functions as defined below:

   * Neutrophils ≥ 1,500 /L
   * Platelets ≥ 100,000 /L
   * Total bilirubin ≤ 1.5 x ULN (upper limit of normal) (except patients with Gilbert's syndrome, who must have a total bilirubin ≤ 3.0 mg/dL)
   * ALT ≤ 2.5 x ULN or ≤ 5 x ULN if liver metastases persist
   * Serum creatinine ≤ 1.5 x ULN or calculated creatinine clearance ≥ 45 mL/minute by the Cockcroft-Gault method
   * Albumin ≥ 3.0 g/dL (≥30 g/L)
   * INR (international normalized ratio) ≤1.4
8. Patients should be able to read and fully understand the requirements of the trial, be willing to comply with all trial visits and assessments, and be willing and able to sign an IRB-approved written informed consent document.
9. Subjects must have recovered from major infections and/or surgical procedures and, in the opinion of the investigator, not have a significant active concurrent medical illness precluding protocol treatment.
10. Patients agree to provide archival tissue block or 10 formalin-fixed paraffin-embedded (FFPE) slides paraffin for use in pharmacodynamics correlative studies.

Exclusion Criteria:

Patients who meet any of the following criteria will be not eligible for the study.

1. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection requiring intravenous antibiotics, symptomatic congestive heart failure (NYHA Class III or IV), or history of myocardial infarction, unstable angina, stroke or transient ischemic attack within 6 months prior to study enrollment.
2. History of clinically significant allergic reactions to the study drugs or their analogs, or any component of the products.
3. Any treatment specific for systemic tumor control within 3 weeks prior to the initiation of the study drugs; or within 2 weeks if cytotoxic agents were given weekly (within 6 weeks for nitrosoureas or mitomycin C), or within 5 half-lives for targeted agents with half-lives and pharmacodynamic effects lasting less than 4 days, or failure to recover from toxic effects of any therapy prior to the study drug treatment.
4. Patients who have not recovered from major surgical procedure, or significant traumatic injury (i.e., still need additional medical care for these issues).
5. History of any of the following cardiovascular events or conditions within the past 6 months prior to enrolment: myocardial infarction, unstable angina, cerebrovascular accident or transient ischemic attack, New York Heart Association Class ≥ II chronic heart failure, significant arrhythmia*; QTcF interval >430 msec or use of drugs that prolong the QT interval at screening; family history of long QT syndrome.

   *Significant arrhythmias are defined as symptoms of syncope or severe palpitations (palpitations requiring referral to cardiac monitoring), or ECG findings of supraventricular tachycardia (including atrial fibrillation or atrial flutter) or ventricular tachycardia (including ventricular fibrillation) or ventricular ectopy (ventricular premature depolarization)
6. Clinically significant and uncontrolled major medical condition(s) that places the subject at an unacceptably high risk for toxicities. These include, but are not limited to: active infections, symptomatic pulmonary disease, inadequate pulmonary function, seizure disorder, or psychiatric illness.
7. Current use of more than one antihypertensive medication.
8. For patients receiving antihypertensive medication: systolic blood pressure <120 mm Hg and/or diastolic blood pressure <70 mm Hg at screening.
9. Major surgical procedure within 4 weeks prior to enrolment.
10. Lactating or pregnant female.
11. Females of childbearing potential and males not using adequate birth control.
12. Current treatment or treatment within 4 weeks of screening with bisphosphonates.
13. Hypocalcemia at screening.
14. History of acute pancreatitis within 6 months prior to screening.
15. Known hypoparathyroidism, pseudohypoparathyroidism, or vitamin D deficiency, or clinical evidence of other conditions known to associated with hypocalcemia, including hypoalbuminemia, hyperphosphatemia, hypomagnesemia.
16. Current treatment or treatment within 4 weeks of screening with drugs known to reduce serum calcium levels, including: bisphosphonates, antiepileptic drugs, cinacalcet, macrolide antibiotics (such as erythromycin, azithromycin), large doses of corticosteroids (>20 mg/day of prednisone or equivalent), or any IV use of corticosteroids. In addition, long-term use (defined as ongoing use for ≥4 weeks) of corticosteroids within 8 weeks of screening is prohibited.
17. Symptomatic and uncontrolled metastasis to the central nervous system or leptomeningeal or lymphangitic carcinomatosis.
18. Grade 2 or higher peripheral neuropathy.
19. Human immunodeficiency virus requiring HAART treatment due to unknown drug-drug interactions or known active hepatitis B or C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events and serious adverse events | Up to 30 days after last dose
  Will assess clinical symptoms and laboratory values, evaluate vital signs and perform physical exams, with a special attention to treatment- related fatigue, gastrointestinal (GI) symptoms, cardiovascular events, myelosuppression, and neurotoxicity.
Incidence of >= grade 2 adverse events according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | Up to 30 days after last dose
Dose-limiting toxicities | Up to 28 days
Withdrawals from the study due to treatment-related adverse events will be documented | Up to 30 days after last dose
Change of the treatment regimen such as dose delay and dose reduction over time by dose level due to treatment-related adverse events | Up to 30 days after last dose

SECONDARY OUTCOMES:
Objective responses | Up to 6 months
  Defined as complete response(CR)s and partial response (PR).
Clinical benefit | Up to 6 months
  Defined as stable disease (SD)/CR/PR according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Predictive biomarkers | Up to 6 months
  Fisher exact test is used to associate potential biomarkers with SD >= 6 months/CR/PR. Next generation sequencing for targeted exome panel and NanoString arrays are used to reveal potential biomarkers of acquired resistance.

CONTACTS AND LOCATIONS:
Overall Officials: Siqing Fu, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org